CLINICAL TRIAL: NCT04426877
Title: Impact Of An Exercise And Nutritional Education Self-Applied Online Intervention On Body Composition And Blood Pressure On Hypertensive Adults With Overweight Or Obesity.
Brief Title: Lifestyle Internet-Based Intervention On Hypertensive Patients With Overweight Or Obesity
Acronym: IBI-HTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-85
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Hypertension; Obesity
Keywords: Hypertension; Obesity; Internet; Exercise; Nutrition
MeSH Terms: conditions — Hypertension; Obesity; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive access to the web-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their hypertension specialist doctor.
  Interventions: Behavioral: Experimental group
- Control Group (Experimental): The control group will receive the same web-based lifestyle intervention (exercise and nutritional education), but in this case supported by audiovisual instructions given by a doctor outside the patient.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Experimental group — The self-applied online program will comprise a three months behavioural intervention composed by 9 modules seeking to develop gradually achieving the goals of changing eating and physical activity habits, supported by audiovisual instructions. This group will receive access to the web-based lifestyle intervention (exercise and nutritional education), supported by audiovisual instructions given by their hypertension specialist doctor.
  Arms: Experimental group
Behavioral: Control group — The self-applied online program will comprise a three months behavioural intervention composed by 9 modules seeking to develop gradually achieving the goals of changing eating and physical activity habits, supported by audiovisual instructions. This group will receive the same web-based lifestyle intervention (exercise and nutritional education), but in this case supported by audiovisual instructions given by a doctor outside the patient.
  Arms: Control Group

SUMMARY:
This study aims to analyze the effects of a 3 months duration self-applied online program, composed of 9 modules focused on promoting healthy lifestyle habits (healthy eating and increased physical activity), on obese or overweight adults with hypertension. Participants will be recruited from a hypertension unit of a public hospital. These patients will be randomized allocated into two interventional groups: experimental group will receive audiovisual instructions from their hypertension specialist doctor, and the control group from a doctor outside the patient. Assessment will include: body composition (BMI), blood pressure, levels of physical activity, functional capacity, fall risk, and quality of life.

DETAILED DESCRIPTION:
Hypertension and obesity or overweight related, even other associated comorbidities, involve a worrying public health problem. The evidence shows that healthy eating and regular physical exercise, monitored by different means (internet, face to face, exercise diaries), play an important prevention role to maintain health while ageing. In this way, Information and Communication Technologies (ICTs) have been demonstrated as a useful tool to promote health, working on barriers at the same time, such as low motivation and difficulties to maintain regular exercise or healthy eating habits. ICTs also allows to reach a wider audience at a lower cost, due to their good cost-benefit relationship and the possibility of increasing the efficiency of interventions. Therefore, this study aims to analyze the effects of a 3 months duration self-applied online program, composed of 9 modules focused on promoting healthy lifestyle habits (healthy eating and increased physical activity), on obese or overweight adults with hypertension. Participants will be recruited from a hypertension unit of a public hospital. These patients will be randomized allocated into two interventional groups: experimental group will receive audiovisual instructions from their hypertension specialist doctor, and the control group from a doctor outside the patient. Assessment will include: body composition (BMI), blood pressure, levels of physical activity, functional capacity, fall risk, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Overweight or obesity (25 ≤ BMI ≤ 35 kg/m2)
* Aged between 18-75 years

Exclusion Criteria:

* Not having access to the Internet or lack of information about it.
* Treatment with more than 3 antihypertensive drugs.
* Meet the criteria of the DSM-IV-TR of a Food Disorder.
* Presenting some type of severe psychiatric disorder.
* Disability that prevents or hinders physical exercise.
* Receiving some treatment for weight loss.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
BMI | At three months
  Body mass index

SECONDARY OUTCOMES:
Blood Pressure (BP) | At three months
  Systolic and diastolic blood pressure
Physical activity | At three months
  Levels of physical activity (measured with SHORT-IPAQ Questionnaire). This Questionnaire measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.
Fall risk | At three months
  Fall risk perception (measured with FES Questionnaire). The 'Falls Efficacy Scale' (FES) directly evaluate the impact of fear of falling on social life. This scale has excellent reliability, is correlated with measures of balance and gait, and predicts future falls and decline in functional capacity. The 16 items of the FES are rated according to "how concerned you are about the possibility of falling", using the following responses (score in parentheses): not at all (1), somewhat (2), fairly (3), and very concerned (4). Thus, the total score ranges from 16 to 64 points. Higher values indicate less fall-related self-efficacy (and more concern about falling).

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L PÁRRAGA, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Enrique Rodilla Sala, Sagunto, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lison JF, Palomar G, Mensorio MS, Banos RM, Cebolla-Marti A, Botella C, Benavent-Caballer V, Rodilla E. Impact of a Web-Based Exercise and Nutritional Education Intervention in Patients Who Are Obese With Hypertension: Randomized Wait-List Controlled Trial. J Med Internet Res. 2020 Apr 14;22(4):e14196. doi: 10.2196/14196. PMID 32286232
- [Derived] Muzquiz-Barbera P, Ruiz-Cortes M, Herrero R, Vara MD, Escriva-Martinez T, Banos RM, Rodilla E, Lison JF. "Own doctor" presence in a web-based lifestyle intervention for adults with obesity and hypertension: A randomized controlled trial. Front Public Health. 2023 Mar 14;11:1115711. doi: 10.3389/fpubh.2023.1115711. eCollection 2023. PMID 36998287